CLINICAL TRIAL: NCT04689971
Title: The Benefits of Vitamin B Combination as Add on Therapy in the Management of Painful Diabetic Neuropathy Patient: Randomized Clinical Trial
Brief Title: The Benefits of Vitamin B Combination as Add on Therapy in the Management of Painful Diabetic Neuropathy Patient
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Duta Wacana Christian University (Other)
Collaborators: PT SOHO Global Health Tbk (Unknown)
Responsible Party: Principal Investigator, Rizaldy Taslim Pinzon, Principal investigator, Neurologist, Duta Wacana Christian University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOHOBION
Record Dates: First submitted 2020-12-19; First posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Painful Diabetic Neuropathy
Keywords: Vitamin B combination; B vitamins; Standard therapy; Diabetic neuropathy; Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Standard of Care; cyanocobalamin, pyridoxine, thiamine drug combination; Vitamin B Complex

STUDY DESIGN:
Intervention Model Description: Eligible subjects were randomly allocated to receive any of the following regiments: standard therapy consists of pregabalin, gabapentine, or amitriptyline (control group) or standard therapy and vitamin B combination (vitamin B1 100 mg, B6 200 mg and B12 200 mcg) tablet once daily (experimental group).
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Receive standard therapy consists of gabapentin, pregabalin, or amitriptyline and vitamin B combination (B1 100 mg, B2 200 mg and B12 200 mcg) tablet once daily (experimental group).
  Interventions: Drug: Standard therapy; Drug: Vitamin B combination
- Control Group (Active Comparator): Receive standard therapy consists of gabapentin, pregabalin, or amitriptyline.
  Interventions: Drug: Standard therapy

INTERVENTIONS:
Drug: Standard therapy — Gabapentin, pregabalin, or amitriptyline
Drug: Vitamin B combination — Vitamin B combination (B1 100 mg, B2 200 mg and B12 200 mcg) tablet once daily
  Other Names: Vitamin B complex
  Arms: Experimental Group

SUMMARY:
Large population-based study has shown that the prevalence of painful diabetic neuropathy (PDN) is around 21%, and painful symptoms are more prevalent in patients with type 2 diabetes, females, and Asians. PDN is characterized by symmetrical lower limb paresthesiae, dysesthesiae, lancinating pains and allodynia, with nocturnal exacerbation. PDN cause sleep disturbance and reduce quality of life. The international guidelines advocate a range of therapies for symptom relief. The therapeutic efficacy for all recommended medications is at best around 50% pain relief and is limited due to unwanted side effects. Apart from peripheral and central alterations, metabolic alterations such as increased glycemic influx, and elevated plasma methylglyoxal levels have been implicated in the pathogenesis of PDN.

Several treatment options for PN are available, including pharmacological, non-pharmacological, and alternative options. Patients suffering from severe and disabling symptoms (e.g. NeP) may require guideline treatments like pregabalin, duloxetine, or gabapentin initially until the symptoms are under control. These medications can symptomatically relieve NeP; however, they do not address the underlying cause. Other options such as neurotropic B vitamins (B1, B6, and B12) do not only target the symptoms, but also improve nerve health and contribute to nerve regeneration. The B vitamins are commonly used for PN treatment in clinical practice worldwide, this treatment option is most suitable before the patient suffers from chronic NeP. However, co-treatment with neurotropic B vitamins is also appropriate in NeP patients, to ensure the restoration of nerve health.

DETAILED DESCRIPTION:
This was randomized clinical trial, active comparator, open label, controlled study from the period of November 2020 - November 2021 at Bethesda Hospital, Yogyakarta, Indonesia.

There were 60 painful diabetic neuropathy patients who fulfilled the inclusion and exclusion criteria. Each subject had been followed up from the first day of medication administration until 8 weeks after medication administration.

Ethical approval number ((kosong)) was obtained from Health Research Ethics Committee, Bethesda Hospital Yogyakarta.

The hypothesis of this study:

a. Add on oral vitamin B combination (B1, B6, and B12) to standard treatment in patients with painful diabetic neuropathy is more effective in reducing pain and neuropathic symptoms in 8 weeks of treatment compared with standard treatment, b. Add on oral vitamin B combination (B1, B6, and B12) to standard treatment in patients with painful diabetic neuropathy is as safe as standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Adult age (>18 years old)
* Diagnosed as painful diabetic neuropathy based on validated Diabetic Neuropathy Symptoms (DNS) and Diabetic Neuropathy Examination (DNE)

Exclusion Criteria:

* Subjects with significant renal and liver problem
* Subjects with known hypersensitivity to vitamin B combination
* Pregnancy and breastfeeding patients
* Patients that enrolled any clinical trial within a month
* Not competent enough in giving approval and answering questionnaires

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-11-03 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Improvement in Visual Analogue Scale (VAS) at week 4 | 4 weeks after treatment initiation
  Change in pain impact on daily life as measured by Visual Analogue Scale (VAS) from its baseline value. Visual analogue scale is a continuous scale comprised of a horizontal or vertical line, usually 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extreme. The scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100). The respondent is asked to place a line perpendicular to the VAS line at the point that represents their pain intensity. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
Improvement in Visual Analogue Scale (VAS) at week 8 | 8 weeks after treatment initiation
  Change in pain impact on daily life as measured by Visual Analogue Scale (VAS) from its baseline and week 4 value. Visual analogue scale is a continuous scale comprised of a horizontal or vertical line, usually 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extreme. The scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100). The respondent is asked to place a line perpendicular to the VAS line at the point that represents their pain intensity. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
Improvement in Numeric Pain Scale at week 4 | 4 weeks after treatment initiation
  Change in pain impact on daily life as measured by Numeric Pain Scale from its baseline value. Numeric pain scale is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. Higher scores indicating greater pain intensity.
Improvement in Numeric Pain Scale at week 8 | 8 weeks after treatment initiation
  Change in pain impact on daily life as measured by Numeric Pain Scale from its baseline and week 4 value. Numeric pain scale is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. Higher scores indicating greater pain intensity.
Improvement in Brief Pain inventory at week 4 | 4 weeks after treatment initiation
  Change in pain impact on daily life as measured by Brief Pain Inventory from its baseline value. The Brief Pain Inventory evaluates a patient's pain experience through a number of different scales. There are line drawings of the front and back of a human body on which patients mark the location of their pain. Patients are asked to list the treatments or medications that they are using and how much relief they have provided in the past 24 hours. In addition, patients fill out 11 different numeric rating scale that ask about pain intensity (ranging from 0 to 10) and the effect of the pain on their ability to function during various activities of daily living. A higher score indicates greater pain intensity.
Improvement in Brief Pain inventory at week 8 | 8 weeks after treatment initiation
  Change in physician global assessment from its baseline value. The Brief Pain Inventory evaluates a patient's pain experience through a number of different scales. There are line drawings of the front and back of a human body on which patients mark the location of their pain. Patients are asked to list the treatments or medications that they are using and how much relief they have provided in the past 24 hours. In addition, patients fill out 11 different numeric rating scale that ask about pain intensity (ranging from 0 to 10) and the effect of the pain on their ability to function during various activities of daily living. A higher score indicates greater pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Rizaldy Pinzon, MD, MSc, PhD, Principal Investigator — Duta Wacana Christian University
Locations (1):
- Bethesda Hospital Yogyakarta, Yogyakarta, Special Region of Yogyakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andres E, Loukili NH, Noel E, Kaltenbach G, Abdelgheni MB, Perrin AE, Noblet-Dick M, Maloisel F, Schlienger JL, Blickle JF. Vitamin B12 (cobalamin) deficiency in elderly patients. CMAJ. 2004 Aug 3;171(3):251-9. doi: 10.1503/cmaj.1031155. PMID 15289425
- [Background] Head KA. Peripheral neuropathy: pathogenic mechanisms and alternative therapies. Altern Med Rev. 2006 Dec;11(4):294-329. PMID 17176168
- [Background] Jayabalan B, Low LL. Vitamin B supplementation for diabetic peripheral neuropathy. Singapore Med J. 2016 Feb;57(2):55-9. doi: 10.11622/smedj.2016027. PMID 26892473
- [Background] Liu KW, Dai LK, Jean W. Metformin-related vitamin B12 deficiency. Age Ageing. 2006 Mar;35(2):200-1. doi: 10.1093/ageing/afj042. PMID 16495296
- [Background] Negrao L, Almeida P, Alcino S, Duro H, Liborio T, Melo Silva U, Figueira R, Goncalves S, Neto Parra L. Effect of the combination of uridine nucleotides, folic acid and vitamin B12 on the clinical expression of peripheral neuropathies. Pain Manag. 2014 May;4(3):191-6. doi: 10.2217/pmt.14.10. Epub 2014 May 16. PMID 24835269
- [Background] Okada K, Tanaka H, Temporin K, Okamoto M, Kuroda Y, Moritomo H, Murase T, Yoshikawa H. Methylcobalamin increases Erk1/2 and Akt activities through the methylation cycle and promotes nerve regeneration in a rat sciatic nerve injury model. Exp Neurol. 2010 Apr;222(2):191-203. doi: 10.1016/j.expneurol.2009.12.017. Epub 2010 Jan 4. PMID 20045411
- [Background] Selvarajah D, Kar D, Khunti K, Davies MJ, Scott AR, Walker J, Tesfaye S. Diabetic peripheral neuropathy: advances in diagnosis and strategies for screening and early intervention. Lancet Diabetes Endocrinol. 2019 Dec;7(12):938-948. doi: 10.1016/S2213-8587(19)30081-6. Epub 2019 Oct 14. PMID 31624024
- [Background] Sun Y, Lai MS, Lu CJ. Effectiveness of vitamin B12 on diabetic neuropathy: systematic review of clinical controlled trials. Acta Neurol Taiwan. 2005 Jun;14(2):48-54. PMID 16008162
- [Background] Tesfaye S, Boulton AJ, Dickenson AH. Mechanisms and management of diabetic painful distal symmetrical polyneuropathy. Diabetes Care. 2013 Sep;36(9):2456-65. doi: 10.2337/dc12-1964. PMID 23970715
- [Background] Ting RZ, Szeto CC, Chan MH, Ma KK, Chow KM. Risk factors of vitamin B(12) deficiency in patients receiving metformin. Arch Intern Med. 2006 Oct 9;166(18):1975-9. doi: 10.1001/archinte.166.18.1975. PMID 17030830